CLINICAL TRIAL: NCT05022706
Title: Accompanying HIV-positive Adolescents Through the Transition Into Adult Care: a Feasibility Study
Brief Title: Pilot Study of a Transition Intervention for ALWH
Acronym: PASEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: University of South Florida (Other); Partners HealthCare (Other); Socios En Salud Sucursal, Peru (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Molly Franke, Associate Professor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB19-0086; 5R21AI143365-02 (NIH)
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Treatment Adherence
Keywords: adolescents; social support; differentiated care; HIV care continuum; key and vulnerable populations
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents living with HIV (Experimental): 1. cART directly observed therapy (DOT) for participants at risk of or with a history of non-adherence
  2. monthly home visits by trained health promoters
  3. ongoing support in navigating the health system, including accompaniment to appointments and assistance enrolling in public health insurance
  4. monthly peer support groups
  Interventions: Other: Community-based accompaniment and home visits; Behavioral: Directly Observed Therapy; Behavioral: Monthly Peer Support Groups

INTERVENTIONS:
Other: Community-based accompaniment and home visits — Trained health promoters will accompany adolescents to their first appointments; facilitate enrollment in public health insurance and completion of other administrative requisites (e.g. obtaining a foreign identification card for migrants; transferring to a different health facility); help troubleshoot new logistical and/or social challenges; and will foster communication between the adult care providers and the patient.
  Health promoters will visit the participant's home or another mutually-agreed upon location at least monthly, to review ART adherence, identify barriers to care and adherence, remind patients of upcoming medical encounters, screen and follow-up for clinical and social problems, and offer social support.
Behavioral: Directly Observed Therapy — Among adolescents who have already initiated combination antiretroviral therapy (cART), directly observed therapy (DOT) will be provided to the subset of adolescents identified as being at high risk of non-adherence, defined by meeting at least one of the following criteria: 1) identified by the pediatric health provider as having unstable adherence; or 2) having a detectable viral load at one of their two previous measurements. In adolescents newly initiating cART, there will not be an adherence precedent. This group will choose whether they wish to receive DOT. As part of this research, trained community health workers (CHWs) will deliver DOT in participant's homes or in a mutually agreed upon location. CHWs will observe ingestion of cART daily, ensure it is taken as prescribed and record each dose as DOT, self-administered, not taken or not prescribed.
Behavioral: Monthly Peer Support Groups — The investigators will assign ALWH to a social support group with 9 to 11 other adolescents also participating in the research. The goal of the social support groups is to provide a venue for participants to share experiences and resources and provide encouragement and support to one another. Each group will last approximately 3 to 4 hours. Support groups will be led by adult peers or trained community health workers. The final group session will incorporate a discussion about the group experience, how it may change behavior, recommendations for improvement, and unmet needs that should be considered for a future intervention.

SUMMARY:
The investigators will conduct a pilot study of a community-based intervention designed to improve outcomes among adolescents living with HIV (ALWH) transitioning to adult HIV care in Lima, Peru. The investigators will enroll adolescents transitioning to adult HIV care, either due to a recent diagnosis or having aged out of their pediatric clinic. ALWH previously lost from care during the transition process will also be invited to participate. The nine-month intervention will consist of (1) logistical, adherence and social support delivered by entry-level health workers who will accompany adolescents during their transition to adult HIV care and (2) group sessions to improve health-related knowledge, skills, and social support. The investigators will assess intervention feasibility and effectiveness in improving medication adherence, psycho-social outcomes, and transition readiness after 6, 9, and 12 months.

DETAILED DESCRIPTION:
Adolescents living with HIV (ALWH) face an elevated risk of poor health outcomes when transitioning into adult-oriented care. Evidence-based interventions to support ALWH during this high-risk period are lacking, especially in Latin America.

The investigators will prospectively enroll adolescents living with HIV into a community-based accompaniment (CBA) intervention to assess the feasibility of the intervention to improve retention with viral load suppression. The intervention will include (a) combined antiretroviral therapy (cART) directly observed therapy (DOT) for participants at risk of or with a history of non-adherence, (b) monthly home visits by trained health promoters to assess adherence and barriers to care and provide social support, (c) ongoing support in navigating the health system, such as accompaniment to appointments and assistance enrolling in public health insurance, and (d) monthly peer support groups. The intervention activities will be delivered more frequently in an intensive phase for 6 months followed by a taper phase for 3 months. The investigators also aim to pilot study procedures relevant to a future trial, including an evaluation of new data collection tools, intervention fidelity assessments, and consent procedures.

Data collection will consist of the use of self-administered questionnaires using RedCap, focus groups with participants, and in-depth interviews with a subset of participants. To examine changes in outcomes throughout the intervention, the investigators will calculate within-person changes from baseline to 6, 9, and 12 months and will use paired t-tests or Wilcoxon signed-rank tests to test whether these quantities differ from zero. The investigators will stratify analyses by early childhood versus recent diagnosis of HIV to understand any differences in effectiveness among subgroups. Data will be analyzed using SAS version 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 21
* HIV-infected and aware of diagnosis
* Currently on or eligible for antiretroviral therapy for HIV, including patients that are lost to treatment follow-up
* Enrolled in HIV care at a participating public sector clinic
* Able to provide informed assent or consent

Exclusion Criteria:

* Living outside of Lima Province

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention: Study refusal rates | Baseline
  The investigators will measure the feasibility of the intervention through acceptability quantitative analyses. These include the study refusal rates (i.e. the proportion of potentially eligible individuals for the study who chose not to participate).
Acceptability and demand of the intervention: Intervention retention rates | 12 months
  The investigators will calculate the intervention retention rates (i.e. the proportion of individuals who were retained in the study) to measure the acceptability and demand of the intervention.
Acceptability of the intervention: Focus groups and in-depth interviews | 10 months, 11 months, and 12 months
  The investigators will also measure the acceptability of the intervention through qualitative analyses including focus groups and in-depth interviews. Focus groups will be conducted with the participants between month 10 and month 12 of their participation in the intervention. These discussions will explore the perception and acceptance of each component of the intervention and potential future adaptations of the study. The in-depth interviews will be carried out to complement and extend the data collected in focus groups. Open-ended questions will be asked to assess 1) how the CBA intervention was perceived and accepted in each group; 2) any adaptations that would need to be made in future studies, and 3) the varying roles of the treatment supporter during the transition.
Demand of the intervention: Group attendance rates | 12 months
  The investigators will assess demand to describe the extent to which the intervention is likely to be used. The investigators will calculate group attendance for study activities. Group attendance will be measured by the proportion of individuals who attended activities, the number of participants who attended at least one session, the median number of groups attended by participants who attended at least one session, the median number of participants per session, and the number of engagements (comments) during virtual sessions.
Evidence of effectiveness of the intervention: combined antiretroviral therapy (cART) adherence | Baseline, 6 months, 9 months, and 12 months
  The investigators will assess the evidence of effectiveness through cART adherence. (i.e. three questions to record self-adherence). The three questions will include, "How many days did you miss at least one dose of any of your ART medications?"; "How often did you take your ART medications correctly?" (5-point scale with 5 representing "always" and 1 representing "never"); and "How well would you say you took your HIV medications, as directed by your doctor?" (6-point scale with 6 representing "excellent" and 1 representing "very bad"). The investigators will calculate the within-person change from baseline to 6, 9, and 12 months to examine changes in outcome and determine if the intervention shows promise of success.
Evidence of effectiveness of the intervention: Psychosocial outcomes | Baseline, 6 months, 9 months, and 12 months
  The investigators will assess the evidence of effectiveness through psychosocial outcomes including self-efficacy, quality of life, and perceived social and instrumental support. These outcomes will be measured using the NIH toolbox (version 2.0) for ages 18-85 on a 5-point ordinal scale ranging from "never" to "always", with higher scores indicating higher levels. The investigators will calculate the within-person change from baseline to 6, 9, and 12 months to examine changes in outcome and determine if the intervention shows promise of success.
Evidence of effectiveness of the intervention: Transition readiness through "Am I on Trac?" | Baseline, 6 months, 9 months, and 12 months
  The investigators will assess transition readiness through "Am I On TRAC?" scales, which consist of knowledge and behavior indices adapted to the local context. The knowledge scale will assess the health condition and general medical self-care of the participant. The behavior scale will measure the frequency with which participants engage in individual health-related behaviors related to transition. The investigators will report the summed score of the subscales. The investigators will calculate the within-person change from baseline to 6, 9, and 12 months to examine changes in outcome and determine if the intervention shows promise of success.
Evidence of effectiveness of the intervention: Transition readiness through Got transition checklist | Baseline, 6 months, 9 months, and 12 months
  The investigators will also assess transition readiness through the "Got Transition?" checklist (version 2.0). This checklist will analyze personal health knowledge and use of medical services. The questionnaire has a 3-point scale ranging from "not my responsibility" to "yes, I know this." The investigators will calculate the within-person change from baseline to 6, 9, and 12 months to examine changes in outcome and determine if the intervention shows promise of success.

CONTACTS AND LOCATIONS:
Overall Officials: Molly F Franke, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (3):
- Peru (3):
  - Hospital Nacional Hipólito Unanue, El Agustino, Lima region
  - Hospital Nacional Arzobispo Loayza, Lima Cercado, Lima region
  - Instituto Nacional de Salud del Nino, San Borja, Lima region

IPD SHARING:
Plan to Share IPD: No
The investigators will not release personal information because the small number of patients consecutively enrolled at each facility, could potentially make them identifiable, even in the absence of direct identifiers